CLINICAL TRIAL: NCT05430399
Title: Utidelone Versus Docetaxel in HER2-negative Locally Advanced or Metastatic Breast Cancer : A Phase III, Open Label, Randomized Controlled Trial
Brief Title: Utidelone Versus Docetaxel in HER2-negative Locally Advanced or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry); Hunan Cancer Hospital (Other)
Responsible Party: Principal Investigator, wang shusen, Chief Physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-2022-UCAN
Record Dates: First submitted 2022-06-02; First posted 2022-06-24 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Breast Neoplasms; Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): utidelone
  Interventions: Drug: utidelone
- Arm B (Active Comparator): docetaxel
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: utidelone — Eligible patients will receive treatment with utidelone(40 mg/ m2 /day, D1-5,Q3W) , treated until disease progression, unacceptable toxicity or patient request for withdrawal, whichever occurs first. Each cycle is 3 weeks in duration.
  Arms: Arm A
Drug: docetaxel — Eligible patients will receive treatment with docetaxel (75mg/ m2/day, D1, Q3W) , treated until disease progression, unacceptable toxicity or patient request for withdrawal, whichever occurs first. Each cycle is 3 weeks in duration.
  Arms: Arm B

SUMMARY:
It is a phase III trial to explore the efficacy and safety of utidelone versus docetaxel in HER2-negative locally advanced or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form;
* Women aged ≥ 18 years;
* Patients with locally advanced or metastatic, histologically or cytologically documented breast cancer;
* The primary tumor and metastases (if re-biopsy was performed) were both HER2-negative;
* Eastern Cooperative Oncology Group (ECOG) score [0-1] points;
* Patients must have metastatic disease that is evaluable on imaging: including at least one measurable lesion (assessed according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1)); or only non-measurable disease as defined by RECIST 1.1 , especially in patients with bone metastases only, while the disease could be documented/assessed by bone scan, PET or MRI;
* Previous chemotherapy with taxane for early breast cancer (eBC; neoadjuvant or adjuvant setting) is permitted if completed ≥12 months before randomization;
* No previous chemotherapy for advanced breast cancer ;
* For HR+ breast cancer patients shall meet one of the two criteria below: a) radiographically confirmed recurrence or progression within 2 years of adjuvant endocrine therapy; b) received at least one line of endocrine therapy in the recurrence or metastasis stage;
* Patients must have recovered to ≤ Grade 1 (CTCAE v5.0) from all toxicities related to prior antineoplastic therapy. However, patients with any grade of alopecia were allowed ;
* Patients with asymptomatic CNS metastases may be enrolled, if:

  1. Intracranial lesions are evaluable and eligible for systemic therapy only in the absence of extracranial evaluable lesions, or
  2. Patients with stable intracranial lesions after local treatment while there are extracranial evaluable lesions ;
* Adequate hematological, hepatic and renal function;
* Women of childbearing potential must agree to use a contraceptive method during the treatment period and for at least 90 days after the last dose of experiment treatment;
* Life expectancy of at least 12 weeks;
* Patients must be able to participate and comply with treatment and follow up.

Exclusion Criteria:

* HER-2 positive (IHC 3+, or FISH positive);
* Other malignancies (including primary brain or leptomeninges-related tumors) within the past 5 years, except cured cutaneous basal cell carcinoma and cervical carcinoma in situ;
* Patients who have received anti-tumor therapy within 4 weeks prior to the start of study treatment, including chemotherapy, radical radiotherapy, biological therapy, immunotherapy or anti-tumor Chinese medicine therapy;
* Patients who have undergone major organ surgery (excluding needle biopsy) or have significant trauma within 4 weeks before the first dose of treatment, or anticipating for a major surgical procedure during the study;
* Experienced grade ≥ 3 nervous system-related adverse events after treatment with anti-microtubule drugs;
* Symptomatic central nervous system metastases;
* Pregnant or lactating women;
* Known or suspected hypersensitivity to any of the study drugs or excipients;
* Any other non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) that precludes study treatment implementation or follow-up ;
* Any other condition that the investigator considers inappropriate to participate in this trial .
* Use of corticosteroids is prohibited.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 60 months
  Time from randomization to progression or death (whichever occurred first)

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 60 months
  The proportion of patients with a best response of CR or PR, according to RECIST 1.1 criteria
Time to response (TTR) | up to 60 months
  the time from randomization to the first documentation of disease response (CR or PR)
Duration of response (DOR) | up to 60 months
  the time from the first evaluation that criteria for CR or PR are met until PD or death is observed, whichever occurs first, calculated only for patients whose best response is evaluated as CR or PR.
Overall survival (OS) | up to 60 months
  Time from randomization to death Time from randomization to death Time from randomization to death Time from randomization to death
Patient-reported health-related quality of life (QoL): FACT-B total score | up to 60 months
  Change from baseline in the FACT-B total score for all questionnaire timepoints. To calculate FACT-B total score patient ratings from 0 (not at all) - 4 (very much) to each of the 37 questionnaire statement are summed up. Total score range: 0 - 148. Higher values indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shusen Wang, Guangzhou, Gangdong
  - Hunan Cancer Hospital, Hunan, Hunan